CLINICAL TRIAL: NCT01409239
Title: Effect of Glycemic Variability on Autonomic Tone in Hospitalized Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kathleen Dungan (Other)
Responsible Party: Sponsor-Investigator, Kathleen Dungan, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTS869
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes; Inpatient
Keywords: hospital; diabetes; glycemic variability; autonomic tone
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous Insulin (Active Comparator)
  Interventions: Drug: Subcutaneous Insulin
- Intravenous insulin (Experimental)
  Interventions: Drug: Intravenous insulin

INTERVENTIONS:
Drug: Intravenous insulin — 24 hr IV insulin administered according to hospital guideline
  Arms: Intravenous insulin
Drug: Subcutaneous Insulin — basal bolus insulin using carb counting technique and insulin analogues
  Arms: Subcutaneous Insulin

SUMMARY:
Glycemic variability has been associated with mortality in hospitalized patients with hyperglycemia. However, it is unknown how modulation of glycemic variability would impact outcomes. One possibility is that glycemic variability could impact autonomic tone. In particular, heart rate variability (HRV) measurement is a sensitive marker for measuring autonomic tone, and aberrations in HRV have been associated with mortality. The current randomized pilot study will compare the effects of continuous intravenous (IV) insulin and subcutaneous basal bolus insulin on glycemic variability and autonomic tone in hospitalized non-critically ill patients with diabetes. Non-critically ill patients who are hyperglycemic or are requiring at least 20 units of insulin per day will be included. Patients with conditions that preclude accurate HRV readings (such as atrial fibrillation or paced rhythms) will be excluded. Patients randomized to intravenous insulin will receive the therapy for 24 hours according to our standard hospital guideline. Patients randomized to subcutaneous (SQ) insulin will receive basal bolus therapy using insulin analogues. All therapies will begin between 8 and 10 AM. Patients will undergo repeated heart rate variability recordings during the 24 hour period. Blood draws will be collected at baseline and at 24 hours for measurement of catecholamines, insulin, and c-peptide. Glycemic variability will be measured using a continuous subcutaneous glucose monitor and reported as coefficient of variation. The primary outcome measure is low frequency-to-high frequency power spectrum ratio of heart rate variability.

1. Glycemic variability is associated with unfavorable changes in autonomic tone, as assessed by low frequency (LF)/high frequency (HF) HRV ratio, independent of changes in overall glycemia.
2. Short-term increases in glycemic variability, followed by more prolonged glycemic stability are observed in generalized hospitalized patients treated with intravenous insulin compared to standardized basal bolus therapy. LF/HF HRV differs among subjects receiving intravenous compared to subcutaneous insulin.
3. Glycemic variability differs among subjects receiving intravenous compared to subcutaneous insulin

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Admitted to a general medicine or medicine subspecialty service
* Insulin use (>20 units/day) or hyperglycemia. Hyperglycemia is defined as glucose greater than 180 mg/dL on at least 2 occasions separated by at least 4 hours apart.

Exclusion Criteria:

* Type 1 diabetes
* Hospital stay expected less than 48 hours
* Inability to consent
* Pregnancy
* Prisoners
* Previous participation
* Autonomic neuropathy
* Conditions that preclude accurate heart rate variability monitoring: atrial fibrillation, frequent ectopy, congestive heart failure, paced heart rhythms
* Conditions which require lower dose insulin algorithms: end stage renal or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Dungan, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from medical wards of the Ohio State University Wexner Medical Center from 9/1/11 to 5/31/12
Pre-assignment Details: Basal insulin was held prior to initiation of IV insulin and all non-insulin diabetes medications were held for the study. 42 patients signed consent. However, 9 subjects were removed due to protocol violation (new arrhythmia 2], new altered mental status [1], initiation of IV insulin [2], early hospital discharge [2], or sensor failure [2].
Groups:
- Subcutaneous Insulin: Among patients receiving subcutaneous insulin, basal and prandial insulin were administered in approximately equal total daily doses with correction dosing. Daily adjustments were based upon 10-20% of the total daily dose.
- Intravenous Insulin: IV insulin was started at 0500 hours the morning following consent. Patients continued to receive prandial and correction insulin until the IV insulin was started, after which only the prandial component was continued. All patients receiving IV insulin were managed using our hospital's universal nursing run guideline, which was adapted from a published protocol and has a target glucose of 6.1-8.3 mmol/l. All floor nurses are trained in its use. Patients were transitioned from the infusion at 1700 hours using approximately 70% of the estimated basal insulin infusion requirement with 4 hours of overlap.
Period: Overall Study
Arm/Group | Subcutaneous Insulin | Intravenous Insulin
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subcutaneous Insulin | Intravenous Insulin | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 15 | 28
  >=65 years | 3 | 2 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (11) | 54 (11) | 54 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 12 | 9 | 21
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Heart Rate Variability Between Intravenous and Subcutaneous Group
Description: difference in mean low frequency/high frequency heart rate variability (LF/HF HRV)at 6 hour. 2 patients were excluded who did not have usable LF/HF HRV data at 6 hours. These patients remained in the study as they did have other measures.
Time Frame: 6 hour
Measure: Median (Inter-Quartile Range); unit: none (ratio)
Arm/Group | Subcutaneous Insulin | Intravenous Insulin
Number analyzed (Participants) | 15 | 16
none (ratio) | 1.0 [0.55 to 2.2] | 2.6 [0.94 to 5.3]
Statistical Analysis 1: Comparison: Subcutaneous Insulin vs Intravenous Insulin; Since this was a pilot study no formal power analysis was possible. It was hypothesized that IV insulin would be associated with lower LF/HF HRV; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney) — Wilcoxon rank-sum was used to determine differences between groups

ADVERSE EVENTS:
Arm/Group | Subcutaneous Insulin | Intravenous Insulin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 3/16 | 1/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous Insulin (N=16) | Intravenous Insulin (N=17)
Hypoglycemia (Endocrine disorders) | 3 (3) | 1 (1) — Hypoglycemia is defined as any glucose <3.9 mmol/l

LIMITATIONS AND CAVEATS:
Since this was a pilot study no formal power analysis was possible. It was hypothesized that IV insulin would be associated with lower LF/HF HRV.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No